CLINICAL TRIAL: NCT02912351
Title: A Post-Market, Single-Center, Retrospective Study to Collect Clinical Outcomes and Safety Data From Patients Who Have Undergone Revision Total Knee Arthroplasty Using Medacta GMK® Revision Prosthesis and Are at Least 2 Years Past Surgery
Brief Title: A Post-Market Retrospective Study on Revision Total Knee Arthroplasty Using Medacta GMK® Revision Prosthesis
Status: Completed | Type: Observational
Sponsor: Medacta USA (Industry)
Responsible Party: Sponsor
Other Study IDs: K102437-01
Record Dates: First submitted 2016-01-04; First posted 2016-09-23 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis
Keywords: Total Knee Arthroplasty; Total Knee Replacement; Revision Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Patient record review, Radiographs, and questionaires. — KSS-Objective Knee Scores, KSS Subsets, Radiographs and Patient Satisfaction

SUMMARY:
This is a retrospective, single-site observational study, designed to assess the clinical outcomes and collect safety data of GMK Revision knee system used for primary or revision total knee arthroplasty at minimum two years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing and able to provide written informed consent for participation in the study. Written informed consent must be obtained prior to any study procedure.
* Patients with ability to understand and provide written authorization for use and disclosure of personal health information
* Patients must be willing to comply with the post-operative evaluation schedule.
* Patients underwent either a primary or revision total knee replacement for any type of etiology (Osteoarthritis, Avascular necrosis, Rheumatoid Arthritis, Post-traumatic Arthritis, Polyarthritis, Primary implantation failure).
* Patients must have received a GMK Revision component
* Patients must be at minimum 2 year (24 months) post-treatment
* The operation was performed or supervised by the investigator.
* No age limit criteria

Exclusion Criteria:

* History of alcoholism
* Currently on chemotherapy or radiation therapy
* Habitual use of narcotic pain medications prior to surgery or after surgery for reasons other than knee pain
* History of a metabolic disorder affecting the skeletal system other than osteoarthritis or osteoporosis
* History of chronic pain issues for reasons other than knee pain
* Women that are pregnant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For patients that had received the treatment modality, GMK Revision Knee System and are at least 2 years (24 months) out from surgery.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-01; Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Total Knee Society Scores (KSS) | Minimum 2 years post surgery
  Total Knee Society Score questionnaire to assess Patient satisfaction and Patient expectations and objective knee scores.

SECONDARY OUTCOMES:
Radiographic Analysis | Minimum 2 years post surgery
  Radiographic analysis will include evaluation of component and limb alignment, evidence of component subsidence or migration and the presence and progression of radiolucent line between the prosthesis, bone and cement.
Patient Satisfaction | Minimum 2 years post surgery
  Assessed with a Likert scale questionnaire for satisfaction of treatment outcome.
Complication Assessment | minimum 2 years post surgery
  by reviewing Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Mukesh Ahuja, MBBS, MS, Study Director — Medacta USA, Inc.
Locations (1):
- Saint Alphonsus Medical Group, Boise, Idaho, United States